CLINICAL TRIAL: NCT01400425
Title: Potential of Florbetapir F 18 PET to Inform Clinical Diagnosis and Management of Patients With Progressive Cognitive Decline
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A17
Record Dates: First submitted 2011-06-09; First posted 2011-07-22 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Progressive Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with Progressive Cognitive Decline (Experimental): Subjects who have previously or are currently being evaluated for progressive cognitive decline. Enrolling physicians must have a confidence of less than 85% in their initial diagnosis of the subject's progressive cognitive decline and that there was at least a 15% chance that the subject's progressive cognitive decline was due to Alzheimer's disease. All subjects who did not complete the study withdrew before receiving a florbetapir F 18 injection and PET scan.
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 370 megabecquerel (MBq) (10 millicurie [mCi]), single dose
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
The study is designed to evaluate whether a florbetapir F 18 PET scan can impact clinical thinking when physicians are determining the likely cause of a subject's cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Are one of the following:

  1. Group A: Recently completed (within the past 18 months) a comprehensive clinical evaluation for progressive cognitive decline.
  2. Group B: Currently being evaluated for progressive cognitive decline with further clinical or laboratory testing still planned.
* Have a site enrolling physician who has

  1. less than high confidence in their diagnosis for the subject related to the cognitive decline at the time of enrollment. The level of confidence in the diagnosis should be rated by the physician as less than 85%, and should be interpreted as the physician estimating that their diagnosis will be correct in less than 85% of patients with the same presentation as the subject; and
  2. suspicion that the subject's cognitive decline is caused, at least in part, by Alzheimer's disease. The level of suspicion should be rated by the physician as there being at least 15% of patients with the same presentation as the subject would have Alzheimer's disease;
* Can tolerate a 10 minute PET scan. The Principal Investigator will carefully assess each subject and use sound medical judgment to determine whether the subject can tolerate the PET scan procedure;
* Have the ability to cooperate and comply with all study procedures;
* Have a study partner willing to accompany the subject on all of the study visits; and
* Give informed consent for study procedures (If the subject is incapable of giving informed consent, the subject's designated decision maker may consent on behalf of the subject but the subject must still confirm assent. This person may serve as the study partner as well).

Exclusion Criteria:

* Subject or site enrolling physician knows the result of a previous amyloid imaging scan.
* Are considered medically unstable;
* Require additional laboratory tests or workup between enrollment and completion of the florbetapir F 18 PET scan;
* Have a clinically significant infectious disease, including Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV) infection;
* Are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days;
* Have ever participated in an experimental study with an amyloid targeting agent unless it can be documented that the subject received only placebo during the course of the trial;
* Have had a radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session; or
* Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception. Females of childbearing potential must not be pregnant (negative serum β-hCG at the time of screening and negative urine β-hCG on the day of imaging) or breast feeding at screening. Females must avoid becoming pregnant, and must agree to refrain from sexual activity or to use reliable contraceptive methods such as prescribed birth control or intrauterine device (IUD) for 24 hours following administration of florbetapir F 18.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (17):
- United States (17):
  - Research Site, Phoenix, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, San Francisco, California
  - Research Site, Boulder, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Shreveport, Louisiana
  - Research Site, Quincy, Massachusetts
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Progressive Cognitive Decline: Subjects who have previously or are currently being evaluated for progressive cognitive decline. Enrolling physicians must have a confidence of less than 85% in their initial diagnosis of the subject's progressive cognitive decline and that there was at least a 15% chance that the subject's progressive cognitive decline was due to Alzheimer's disease. All subjects who did not complete the study withdrew before receiving a florbetapir F 18 injection and PET scan. Subjects received IV injection, 370 MBq (10 mCi) florbetapir F18, single dose.
Period: Overall Study
Arm/Group | Subjects With Progressive Cognitive Decline
Started | 239
Completed | 229
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Progressive Cognitive Decline
Number analyzed (Participants) | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 205
Age Continuous [Mean (Standard Deviation); unit: years] | 74.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 115
Region of Enrollment [Number; unit: participants]
  United States | 229

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Undergo a Hypothetical Change in Clinical Diagnosis and Physician Management Plan After Obtaining a Negative Florbetapir F 18 PET Scan.
Description: The impact of a negative florbetapir F 18 PET scan on a physician's clinical diagnosis and management of a subject was evaluated on a hypothetical basis because at the start of this study Florbetapir F 18 was an investigational drug and the data collected is for research purposes only. The percentage of subjects who received a negative florbetapir scan that led to a change in hypothetical clinical diagnosis and physician management plans are presented below. A negative florbetapir PET scan is indicative of none to sparse β-amyloid neuritic plaque density according to the modified Consortium to Establish a Registry for Alzheimer's Disease (CERAD) criteria.
Time Frame: 6 weeks
Population: 116 of 229 subjects with progressive cognitive decline received a negative florbetapir scan.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Subjects With Progressive Cognitive Decline
Number analyzed (Participants) | 116
Percentage of subjects
  Change in Clinical Diagnosis | 56.9 [47.8 to 65.5]
  Change in Physician Management Plan | 81.9 [73.9 to 87.8]

2. Secondary Outcome: Percentage of Subjects Who Undergo a Hypothetical Change in Clinical Diagnosis and Physician Management Plan After Obtaining a Positive Florbetapir F 18 PET Scan
Description: The impact of a positive florbetapir F 18 PET scan on a physician's clinical diagnosis and management of a subject was evaluated on a hypothetical basis because at the start of this study Florbetapir F 18 was an investigational drug and the data collected is for research purposes only. The percentage of subjects who received a positive florbetapir scan that led to a change in hypothetical clinical diagnosis and physician management plans are presented below. A positive florbetapir PET scan is indicative of moderate to frequent β-amyloid neuritic plaque density according to the modified Consortium to Establish a Registry for Alzheimer's Disease (CERAD) criteria.
Time Frame: 6 weeks
Population: 113 out of 229 subjects with progressive cognitive decline received a positive florbetapir scan.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Subjects With Progressive Cognitive Decline
Number analyzed (Participants) | 113
Percentage of subjects
  Change in Clinical Diagnosis | 52.2 [43.1 to 61.2]
  Change in Physician Management Plan | 92.0 [85.6 to 95.8]

3. Other Pre Specified Outcome: Item Wise Changes in Physician Management Plan
Description: This outcome analyzed the percentage of subjects who had a hypothetical change in one of the medication or diagnostic categories listed below after receiving a florbetapir scan.
Time Frame: 6 weeks
Population: The number of subjects analyzed for each reporting group is determined by scan status. There were 229 total subjects with progressive cognitive decline of whom 113 received a positive florbetapir scan and 116 received a negative florbetapir scan.
Measure: Number; unit: Percentage of subjects
Groups:
- Subjectss With a Positive Scan: Subjects with progressive cognitive decline that received a positive florbetapir scan.
- Subjects With a Negative Scan: Subjects with progressive cognitive decline that received a negative scan.
Arm/Group | Subjects With Progressive Cognitive Decline | Subjectss With a Positive Scan | Subjects With a Negative Scan
Number analyzed (Participants) | 229 | 113 | 116
Percentage of subjects
  AD Medication | 31.0 | 31.9 | 30.2
  Psychiatric Medication | 7.4 | 3.5 | 11.2
  Refer to Clinical Trial | 16.2 | 22.1 | 10.3
  Brain Structural Imaging (CT/MRI) | 14.0 | 15.0 | 12.9
  Lumbar Puncture | 10.5 | 8.8 | 12.1
  Neuropsychologic Testing | 22.7 | 23.9 | 21.6
  FDG PET | 10.0 | 10.6 | 9.5
  ApoE Genotype | 5.2 | 5.3 | 5.2
  Lab Test | 7.9 | 10.6 | 5.2

4. Secondary Outcome: Change in Confidence of the Clinical Diagnosis
Description: Change in confidence of the clinical diagnosis prior to obtaining a florbetapir F 18 PET scan to the confidence after obtaining a florbetapir F 18 PET scan among subjects in whom the clinical diagnosis remains unchanged. Confidence levels were self-determined by physicians based on their diagnostic certainty and ranged from 0-100%. The mean (SD) change in confidence reflects the average change in diagnostic confidence along the 0-100% scale for the 62 subjects analyzed.
Time Frame: 6 weeks
Population: The hypothetical clinical diagnosis remained unchanged in 62 of 229 subjects who received a florbetapir scan.
Measure: Mean (Standard Deviation); unit: Percent Change in Confidence
Arm/Group | Subjects With Progressive Cognitive Decline
Number analyzed (Participants) | 62
Percent Change in Confidence | 23 (11.9)

5. Secondary Outcome: Change in Physician Management Plans
Description: Determine the percentage of subjects that had at least one hypothetical change between pre and post scan physician management plans. Change in management is defined as the number of subjects prescribed different item-wise plans at the two assessments divided by the total number of subjects in the population with both a pre and post florbetapir F 18 PET scan physician management plan.
Time Frame: 6 weeks
Population: All subjects with progressive cognitive decline who have received a florbetapir scan.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Subjects With Progressive Cognitive Decline
Number analyzed (Participants) | 229
Percentage of subjects | 86.9 [81.9 to 90.7]

6. Other Pre Specified Outcome: Percentage of Subjects Who Undergo a Hypothetical Change in Clinical Diagnosis After Obtaining a Florbetapir F 18 PET Scan.
Description: The impact of a florbetapir F 18 PET scan on a physician's clinical diagnosis of a subject was evaluated on a hypothetical basis because at the start of this study Florbetapir F 18 was an investigational drug and the data collected is for research purposes only. The percentage of subjects who received a florbetapir scan that led to a change in hypothetical clinical diagnosis is presented below.
Time Frame: 6 weeks
Population: Subjects who have received a florbetapir scan (either positive or negative).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Subjects With Progressive Cognitive Decline
Number analyzed (Participants) | 229
Percentage of subjects | 54.6 [48.1 to 60.9]

ADVERSE EVENTS:
Arm/Group | Subjects With Progressive Cognitive Decline
Serious Adverse Events (participants affected / at risk) | 0/229
Other Adverse Events (participants affected / at risk) | 13/229
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Progressive Cognitive Decline (N=229)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Balance disorder (Nervous system disorders) | 1 (1)
Crying (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less